CLINICAL TRIAL: NCT04261491
Title: Impact of Scaling and Root Planing on Systemic Inflammation and Serum Bone Resorption Markers in Postmenopausal Women With Low Bone Mineral Density With Periodontitis.
Brief Title: Impact of SRP on Bone Resorption and Systemic Inflammatory Markers in Postmenopausal Women With Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: roma rathee perio
Record Dates: First submitted 2020-02-03; First posted 2020-02-07 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Tooth Exfoliation; Root Planing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- postmenopausal women with chronic periodontitis (Experimental): postmenopausal women with chronic periodontitis will be evaluated after SRP for serum bone resorption markers- CTX and inflammatory markers IL-6
  Interventions: Procedure: scaling and root planing

INTERVENTIONS:
Procedure: scaling and root planing — scaling and root planing

SUMMARY:
This study is designed to determine the effect of treating postmenopausal women and using non-surgical techniques on biomarkers of systemic inflammation (IL-6 ) and systemic bone resorption (C-terminal collagen cross-links, CTX).

DETAILED DESCRIPTION:
Periodontitis is an inflammatory disease of tooth supporting tissues that is characterized by progressive loss of bone and periodontal attachment and which ultimately leads to tooth loss if left untreated. It is a widespread condition which affects 30% of the adult population. The prevalence increases to greater than 47% among adults age 30 years or older, with those over 65 years old accounting for most cases Osteoporosis is a disease characterized by low bone mineral density(BMD) and deterioration of bone microarchitecture, which leads to increased risk of fragility fractures. It has been reported that one out of two Indian females above the age of 50 years and one out of five Indian men above the age of 65 years are at risk of osteoporosis. It is apparent that both periodontitis and osteoporosis are chronic conditions characterized by resorptive osseous changes with multiple shared risk factors including age, genetics, hormonal change, smoking , as well as calcium and vitamin D deficiency. It has been proposed that the two diseases could also have a mutual relation and this has led to a considerable number of studies investigating the same .Both osteoporosis and periodontitis are more prevalent among elderly population. The number of patients who suffer from both periodontitis and osteoporosis is expected to rise as the average lifespan increases.

Eighty percent of individuals with osteoporosis are women, largely due to the marked loss in bone density associated with the withdrawal of estrogen that accompanies loss of ovarian function at menopause. There is now strong evidence to suggest that systemic pro-inflammatory cytokines in response to estrogen withdrawal at menopause is responsible for increased osteoclastic activity.Systemic Inflammation results in an uncoupling between bone resorption and formation and favours excessive bone resorption resulting in decreased bone mineral density and increased fracture risk in postmenopausal women. Pro-inflammatory cytokines capable of stimulating osteoclastic bone resorption include IL-1, TNF-α, IL-6,IL-11, IL-15 and IL-17. It has been demonstrated that while periodontitis is a local infectious disease of tooth supporting structures, it is also associated with higher inflammatory mediators in the systemic circulation. The data suggest that an individual's overall bone metabolism might be associated with periodontal disease and be reflective of its progression.

Levels of bone turnover markers (BTM) reflect the activity and number of bone forming (osteoblasts) and bone-degrading (osteoclasts) cells, providing an estimate of bone resorption and bone formation. BTM can be measured non-invasively in either blood or urine at a fairly low cost. C-terminal collagen cross-links,CTX, is a bone resorption marker which consists of cross-linked telopeptides from collagen which are released during enzymatic degradation of bone matrix by the osteoclasts Scaling and root planing (SRP) is the most accepted treatment for managing chronic periodontitis and is proven to be effective at controlling local inflammation. Recent research has found evidence that levels of systemic inflammatory markers including IL-1, TNF-α, and IL-6 are also reduced after SRP. Therefore, treatment of periodontal disease results in reduced systemic inflammation but it is unknown if this translates to better outcomes for management of osteoporosis. It is hypothesized that if periodontitis has an influence on bone remodeling, then levels of BTM would also vary with decrease in systemic inflammation owing to resolution of periodontal inflammation following non-surgical periodontal treatment. The purpose of this study is to determine the effect of treating periodontal disease in patients with osteoporosis with scaling and root planing on biomarkers of systemic inflammation (IL-6) and systemic bone turnover (CTX). It is anticipated that the results of this study could be useful in formulating recommendations for interdisciplinary management of patients of concomitant periodontitis and osteoporosis.

MATERIALS AND METHODOLOGY

STUDY DESIGN SETTING: The present prospective interventional study will be conducted in department of Periodontology , Post Graduate institute Dental Sciences,Rohtak.

STUDY PERIOD: 14 months STUDY POPULATION : Patients will be recruited from out patient department of Periodontology.

METHODOLOGY The study will be conducted as follows .

METHOD OF RECRUITMENT:

Post-menopausal females diagnosed with stage 2 and stage 3 periodontitis will be recruited from the outpatient department of Periodontology. Only those patients who consent for the study will be included after obtaining an informed written consent. Those who fulfill the inclusion criteria will be enrolled in the study. Clinical periodontal parameters (CAL, PD and BOP) will be recorded and venous blood samples for measuring serum levels of IL-6 and sCTX will be collected. Scaling and root planing will be performed in all cases. All patients will be re-evaluated after 8 weeks for recording clinical periodontal parameters and serum inflammatory and bone resorption markers as before.

INTERVENTION Full mouth scaling and root planing (SRP) will be performed for all participants with both ultrasonic instruments and manual instrumentation using scalers and curettes. All patients will be given instructions for maintaining proper oral hygiene using soft toothbrush and fluoridated toothpaste. No mouthwashes will be prescribed.

FOLLOW UP OF STUDY PARTICIPANTS All participants will be evaluated for clinical periodontal parameters (PD, CAL and BOP) at 8 weeks after completion of SRP. Serum inflammatory (IL-6) and bone resorption markers (CTX) will be evaluated only for those participants in whom <10 % bleeding sites .

BODY MASS INDEX (BMI) BMI=Weight(kg)/Height²(m²)

BIOCHEMICAL PARAMETERS Venous blood from the anticubital vein will be collected after overnight fasting after applying a tourniquet in a plain vacutainer tube without additive. Immediately after collection of blood samples,the samples will be centrifuged, and separated serum and plasma will be stored at -80̊ c until processed. The level of following biomarkers will be evaluated using ELISA kits- IL-6,sCTX All the blood samples will be collected at the baseline and 8 weeks following SRP.

ELIGIBILITY:
Inclusion Criteria-

* Females in natural menopause since at least 5 years
* Periodontitis with 20 or more natural teeth (excluding third molars). Periodontitis criteria
* Periodontal classification stage 2 or stage 3 (2017 World Workshop on Classification of Periodontal and Peri-Implant Diseases and Conditions)
* More than 30% of sites bleeding on probing. Exclusion Criteria
* Systemic disease known to effect BMD including rheumatoid arthritis, ankylosing spondylitis, and chronic obstructive pulmonary disease.
* Systemic disease known to aﬀect the course of periodontal disease like diabetes mellitus or immunologic disorders
* Treatment with the following drugs in the previous 3 months: steroids, immune suppressants, antibiotics, anti-inﬂammatory drugs, statins, anti-convulsants, thiazide diuretic agents, anti-coagulants, or any other host modulatory drugs
* Recent history or presence of acute or chronic infection.
* History of metabolic bone disease, thyroid and parathyroid disease, and gastrointestinal disorders
* Early onset of menopause
* Treatment for low BMD with systemic medication including calcium and vitamin D supplementation, bisphosphonates, and hormone replacement therapy
* History of hysterectomy
* Current or former smokers or use of smokeless tobacco in any form
* periodontal treatment within 1 year prior to inclusion into the study

Ages: 52 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 52-70 years of females with Chronic Periodontitis
Enrollment: 38 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
serum IL-6, | 2 months
  change in serum IL-6,
s-CTX | 2 months
  change in serum carboxy terminal collagen cross links

SECONDARY OUTCOMES:
Platelet count | 2 months
  change in platelet count
platelet distribution width PDW | 2 months
  change in platelet distribution width PDW
mean platalet volume | 2 months
  change in mean platelet volume

CONTACTS AND LOCATIONS:
Overall Officials: ROMA RATHEE, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCES
Locations (2):
- India (2):
  - Post Graduate Institute of Dental Sciences, Rohtak, Haryana
  - Sanjay Tewari, Rohtak, Haryana

IPD SHARING:
Plan to Share IPD: Yes
study protocol
Supporting Information: Study Protocol